CLINICAL TRIAL: NCT01078090
Title: Effectiveness and Safety of Adalimumab in Rheumatoid Arthritis Patients in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: HUM 03-1
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Safety; Rheumatoid Arthritis; Effectiveness
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid arthritis: Participants with rheumatoid arthritis prescribed adalimumab in routine clinical practice were observed from the first dose for up to 5 years.

SUMMARY:
Observation of safety, tolerability and effectiveness of adalimumab (Humira) therapy in a large patient collective under everyday clinical conditions over a 5-year period.

DETAILED DESCRIPTION:
Patients with Rheumatoid Arthritis and started treatment with adalimumab in a normal clinical setting according to the label were documented. The follow-up observation period was for 5 years and focused on safety information and maintenance of efficacy during the normal clinical setting. Follow-up with participants was via regular office visits at intervals as determined by routine clinical practice or as recommended by national guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe active rheumatoid arthritis in adults with insufficient response to disease-modifying antirheumatic drugs, including methotrexate.
* Moderate to severe active rheumatoid arthritis in adults who have not been treated with methotrexate before.
* In case of incompatibility with methotrexate, adalimumab can be used as monotherapy

Exclusion Criteria:

* Hypersensitivity against the drug or one of the other ingredients; active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections); moderate to severe cardiac insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population: patients with rheumatoid arthritis who resided in Germany. German regulations state that all patients are eligible for non-interventional studies; there are no exclusions. Adult patients (≥ 18 years of age) with RA who were preparing to initiate adalimumab therapy according to the product label were eligible for study enrollment. The eligibility criteria below reflect the approved label as stated in the German Summary of Product Characteristics (SPC) for Humira.
Sampling Method: Non-Probability Sample
Enrollment: 5745 (Actual)
Dates: Start 2003-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Wittig, MD, Study Director — AbbVie Deutschland GmbH & Co. KG, Medical Department
Locations (370):
- Germany (370):
  - Site Reference ID/Investigator# 35034, Aachen
  - Site Reference ID/Investigator# 35033, Aachen
  - Site Reference ID/Investigator# 53919, Achern
  - Site Reference ID/Investigator# 53883, Aichhalden
  - Site Reference ID/Investigator# 35041, Altenburg
  - Site Reference ID/Investigator# 35050, Amberg
  - Site Reference ID/Investigator# 53974, Amberg
  - Site Reference ID/Investigator# 33347, Augsburg
  - Site Reference ID/Investigator# 33356, Bad Abbach
  - Site Reference ID/Investigator# 33359, Bad Abbach
  - Site Reference ID/Investigator# 33362, Bad Aibling
  - Site Reference ID/Investigator# 35084, Bad Aibling
  - Site Reference ID/Investigator# 53968, Bad Aibling
  - Site Reference ID/Investigator# 53966, Bad Bellingen
  - Site Reference ID/Investigator# 35523, Bad Bentheim
  - Site Reference ID/Investigator# 35571, Bad Bramstedt
  - Site Reference ID/Investigator# 53903, Bad Bramstedt
  - Site Reference ID/Investigator# 53929, Bad Buchau
  - Site Reference ID/Investigator# 33370, Bad Endbach
  - Site Reference ID/Investigator# 33369, Bad Endbach
  - Site Reference ID/Investigator# 33380, Bad Iburg
  - Site Reference ID/Investigator# 33384, Bad Kissingen
  - Site Reference ID/Investigator# 33385, Bad Kreuznach
  - Site Reference ID/Investigator# 33389, Bad Liebenwerda
  - Site Reference ID/Investigator# 53942, Bad Mergentheim
  - Site Reference ID/Investigator# 33394, Bad Münder am Deister
  - Site Reference ID/Investigator# 33398, Bad Nauheim
  - Site Reference ID/Investigator# 33399, Bad Neuenahr
  - Site Reference ID/Investigator# 35576, Bad Neuenahr
  - Site Reference ID/Investigator# 53980, Bad Pyrmont
  - Site Reference ID/Investigator# 33402, Bad Rappenau
  - Site Reference ID/Investigator# 33410, Bad Soden-Salmünster
  - Site Reference ID/Investigator# 33415, Bad Staffelstein
  - Site Reference ID/Investigator# 54804, Bad Tölz
  - Site Reference ID/Investigator# 33423, Baden-Baden
  - Site Reference ID/Investigator# 33427, Bamberg
  - Site Reference ID/Investigator# 33436, Bautzen
  - Site Reference ID/Investigator# 33440, Bayreuth
  - Site Reference ID/Investigator# 53978, Belm
  - Site Reference ID/Investigator# 33449, Bensheim
  - Site Reference ID/Investigator# 33646, Berlin
  - Site Reference ID/Investigator# 53902, Berlin
  - Site Reference ID/Investigator# 33662, Berlin
  - Site Reference ID/Investigator# 33695, Berlin
  - Site Reference ID/Investigator# 34243, Berlin
  - Site Reference ID/Investigator# 33681, Berlin
  - Site Reference ID/Investigator# 35599, Berlin
  - Site Reference ID/Investigator# 53959, Berlin
  - Site Reference ID/Investigator# 33688, Berlin
  - Site Reference ID/Investigator# 34260, Berlin
  - Site Reference ID/Investigator# 33685, Berlin
  - Site Reference ID/Investigator# 53948, Berlin
  - Site Reference ID/Investigator# 53939, Berlin
  - Site Reference ID/Investigator# 53971, Berlin
  - Site Reference ID/Investigator# 53933, Berlin
  - Site Reference ID/Investigator# 53884, Berlin
  - Site Reference ID/Investigator# 33672, Berlin
  - Site Reference ID/Investigator# 35552, Berlin
  - Site Reference ID/Investigator# 35554, Bernau
  - Site Reference ID/Investigator# 53899, Biberach
  - Site Reference ID/Investigator# 34279, Bielefeld
  - Site Reference ID/Investigator# 54810, Bielefeld
  - Site Reference ID/Investigator# 35559, Bietigheim-Bissingen
  - Site Reference ID/Investigator# 35560, Bietigheim-Bissingen
  - Site Reference ID/Investigator# 34283, Blankenburg/Hart
  - Site Reference ID/Investigator# 34286, Blaubeuren Abbey
  - Site Reference ID/Investigator# 34289, Bocholt
  - Site Reference ID/Investigator# 53946, Bocholt
  - Site Reference ID/Investigator# 35567, Bochum
  - Site Reference ID/Investigator# 35642, Bogen
  - Site Reference ID/Investigator# 34300, Bonn
  - Site Reference ID/Investigator# 53969, Bonn
  - Site Reference ID/Investigator# 35647, Bonn
  - Site Reference ID/Investigator# 35648, Bonn
  - Site Reference ID/Investigator# 34294, Bonn
  - Site Reference ID/Investigator# 34305, Braunschweig
  - Site Reference ID/Investigator# 34310, Braunschweig
  - Site Reference ID/Investigator# 35601, Breitenbrunn
  - Site Reference ID/Investigator# 35607, Bremen
  - Site Reference ID/Investigator# 53975, Bremen
  - Site Reference ID/Investigator# 34264, Buch
  - Site Reference ID/Investigator# 53934, Büchen
  - Site Reference ID/Investigator# 34696, Celle
  - Site Reference ID/Investigator# 34700, Chemnitz
  - Site Reference ID/Investigator# 35092, Chemnitz
  - Site Reference ID/Investigator# 33990, Cologne
  - Site Reference ID/Investigator# 33987, Cologne
  - Site Reference ID/Investigator# 33996, Cologne
  - Site Reference ID/Investigator# 33993, Cologne
  - Site Reference ID/Investigator# 35238, Cologne
  - Site Reference ID/Investigator# 35617, Cottbus
  - Site Reference ID/Investigator# 53987, Cuxhaven
  - Site Reference ID/Investigator# 53889, Cuxhaven
  - Site Reference ID/Investigator# 35622, Darmstadt
  - Site Reference ID/Investigator# 53885, Delmenhorst
  - Site Reference ID/Investigator# 34726, Demmin
  - Site Reference ID/Investigator# 53932, Denkendorf
  - Site Reference ID/Investigator# 35636, Dortmund
  - Site Reference ID/Investigator# 35632, Dortmund
  - Site Reference ID/Investigator# 35171, Dresden
  - Site Reference ID/Investigator# 34762, Dresden
  - Site Reference ID/Investigator# 53958, Dresden
  - Site Reference ID/Investigator# 34749, Dresden
  - Site Reference ID/Investigator# 34763, Dresden
  - Site Reference ID/Investigator# 34776, Duisburg
  - Site Reference ID/Investigator# 53897, Duisburg
  - Site Reference ID/Investigator# 34771, Düsseldorf
  - Site Reference ID/Investigator# 34774, Düsseldorf
  - Site Reference ID/Investigator# 34779, Ebensfeld
  - Site Reference ID/Investigator# 34782, Eberswalde
  - Site Reference ID/Investigator# 54805, Eisenberg
  - Site Reference ID/Investigator# 35180, Elmshorn
  - Site Reference ID/Investigator# 34802, Erftstadt
  - Site Reference ID/Investigator# 34807, Erfurt
  - Site Reference ID/Investigator# 35097, Erfurt
  - Site Reference ID/Investigator# 35189, Erfurt
  - Site Reference ID/Investigator# 54811, Erlangen
  - Site Reference ID/Investigator# 34815, Erlangen
  - Site Reference ID/Investigator# 53925, Essen
  - Site Reference ID/Investigator# 34823, Essen
  - Site Reference ID/Investigator# 35194, Essen
  - Site Reference ID/Investigator# 53931, Essen
  - Site Reference ID/Investigator# 53945, Essen
  - Site Reference ID/Investigator# 34829, Esslingen am Neckar
  - Site Reference ID/Investigator# 35200, Feldafing
  - Site Reference ID/Investigator# 35203, Flensburg
  - Site Reference ID/Investigator# 34831, Forchheim
  - Site Reference ID/Investigator# 34851, Frankfurt
  - Site Reference ID/Investigator# 34838, Frankfurt
  - Site Reference ID/Investigator# 35211, Fraureuth
  - Site Reference ID/Investigator# 35217, Freiberg
  - Site Reference ID/Investigator# 34852, Freiburg im Breisgau
  - Site Reference ID/Investigator# 34855, Freiburg im Breisgau
  - Site Reference ID/Investigator# 53926, Freiburg im Breisgau
  - Site Reference ID/Investigator# 34859, Freiburg im Breisgau
  - Site Reference ID/Investigator# 35099, Freystadt
  - Site Reference ID/Investigator# 53960, Friedberg
  - Site Reference ID/Investigator# 35222, Friedrichroda
  - Site Reference ID/Investigator# 53976, Geesthacht
  - Site Reference ID/Investigator# 53890, Geilenkirchen
  - Site Reference ID/Investigator# 34877, Gelsenkirchen
  - Site Reference ID/Investigator# 53909, Giessen
  - Site Reference ID/Investigator# 53922, Gladbeck
  - Site Reference ID/Investigator# 34894, Goslar
  - Site Reference ID/Investigator# 35231, Göttingen
  - Site Reference ID/Investigator# 65622, Göttingen
  - Site Reference ID/Investigator# 34902, Greifswald
  - Site Reference ID/Investigator# 53957, Groß Reken
  - Site Reference ID/Investigator# 34910, Güstrow
  - Site Reference ID/Investigator# 35501, Hagen
  - Site Reference ID/Investigator# 34924, Halle
  - Site Reference ID/Investigator# 34935, Halle
  - Site Reference ID/Investigator# 34938, Halle
  - Site Reference ID/Investigator# 34920, Halle
  - Site Reference ID/Investigator# 34942, Halle
  - Site Reference ID/Investigator# 33819, Halle
  - Site Reference ID/Investigator# 35442, Hamburg
  - Site Reference ID/Investigator# 53984, Hamburg
  - Site Reference ID/Investigator# 33367, Hamburg
  - Site Reference ID/Investigator# 53900, Hamburg
  - Site Reference ID/Investigator# 34956, Hamburg
  - Site Reference ID/Investigator# 34962, Hamburg
  - Site Reference ID/Investigator# 35450, Hamburg
  - Site Reference ID/Investigator# 35112, Hamburg
  - Site Reference ID/Investigator# 34946, Hamburg
  - Site Reference ID/Investigator# 35001, Hamburg
  - Site Reference ID/Investigator# 34959, Hamburg
  - Site Reference ID/Investigator# 34977, Hamburg
  - Site Reference ID/Investigator# 34965, Hamburg
  - Site Reference ID/Investigator# 54806, Hamburg
  - Site Reference ID/Investigator# 33578, Hamburg
  - Site Reference ID/Investigator# 34967, Hamburg
  - Site Reference ID/Investigator# 34989, Hamburg
  - Site Reference ID/Investigator# 34981, Hamburg
  - Site Reference ID/Investigator# 34984, Hamburg
  - Site Reference ID/Investigator# 34996, Hamburg
  - Site Reference ID/Investigator# 53953, Hamm
  - Site Reference ID/Investigator# 35017, Hanau
  - Site Reference ID/Investigator# 33713, Hanover
  - Site Reference ID/Investigator# 35032, Hanover
  - Site Reference ID/Investigator# 35021, Hanover
  - Site Reference ID/Investigator# 33788, Hanover
  - Site Reference ID/Investigator# 33790, Harrislee
  - Site Reference ID/Investigator# 65629, Haselünne
  - Site Reference ID/Investigator# 33795, Hattingen
  - Site Reference ID/Investigator# 33796, Heidelberg
  - Site Reference ID/Investigator# 33806, Heidelberg
  - Site Reference ID/Investigator# 33811, Heidelberg
  - Site Reference ID/Investigator# 33816, Heilbad Heiligenstadt
  - Site Reference ID/Investigator# 53911, Herne
  - Site Reference ID/Investigator# 53910, Herne
  - Site Reference ID/Investigator# 65623, Herne
  - Site Reference ID/Investigator# 33823, Herrsching am Ammersee
  - Site Reference ID/Investigator# 33831, Hildesheim
  - Site Reference ID/Investigator# 33836, Hof
  - Site Reference ID/Investigator# 33840, Hofheim
  - Site Reference ID/Investigator# 33843, Hohenfelde
  - Site Reference ID/Investigator# 54807, Homburg
  - Site Reference ID/Investigator# 53985, Illingen
  - Site Reference ID/Investigator# 33933, Ingolstadt
  - Site Reference ID/Investigator# 53938, Jena
  - Site Reference ID/Investigator# 5323, Jena
  - Site Reference ID/Investigator# 33940, Jülich
  - Site Reference ID/Investigator# 33944, Kahla
  - Site Reference ID/Investigator# 35124, Kahla
  - Site Reference ID/Investigator# 33948, Kaiserslautern
  - Site Reference ID/Investigator# 53935, Kaltenkirchen
  - Site Reference ID/Investigator# 33397, Karlsruhe
  - Site Reference ID/Investigator# 33954, Karlsruhe
  - Site Reference ID/Investigator# 35482, Karlstadt am Main
  - Site Reference ID/Investigator# 33962, Kassel
  - Site Reference ID/Investigator# 35239, Kolkwitz
  - Site Reference ID/Investigator# 34000, Königs Wusterhausen
  - Site Reference ID/Investigator# 34006, Kressbronn
  - Site Reference ID/Investigator# 34009, Kronach
  - Site Reference ID/Investigator# 34086, Kyritz
  - Site Reference ID/Investigator# 34003, Lahr
  - Site Reference ID/Investigator# 53937, Leipzig
  - Site Reference ID/Investigator# 65628, Leipzig
  - Site Reference ID/Investigator# 34107, Leipzig
  - Site Reference ID/Investigator# 34098, Leipzig
  - Site Reference ID/Investigator# 34119, Leverkusen
  - Site Reference ID/Investigator# 34121, Lichtenstein
  - Site Reference ID/Investigator# 35252, Lippstadt
  - Site Reference ID/Investigator# 53882, Löhne
  - Site Reference ID/Investigator# 53886, Ludwigsburg
  - Site Reference ID/Investigator# 35257, Ludwigsfelde
  - Site Reference ID/Investigator# 53906, Ludwigslust
  - Site Reference ID/Investigator# 34133, Lübeck
  - Site Reference ID/Investigator# 53943, Lüdenscheid
  - Site Reference ID/Investigator# 33407, Lüneburg
  - Site Reference ID/Investigator# 53888, Lüneburg
  - Site Reference ID/Investigator# 34148, Magdeburg
  - Site Reference ID/Investigator# 53981, Magdeburg
  - Site Reference ID/Investigator# 53913, Magdeburg
  - Site Reference ID/Investigator# 53928, Mainz
  - Site Reference ID/Investigator# 65631, Mainz
  - Site Reference ID/Investigator# 34184, Mannheim
  - Site Reference ID/Investigator# 34194, Marl
  - Site Reference ID/Investigator# 35283, Menz
  - Site Reference ID/Investigator# 53896, Merxheim
  - Site Reference ID/Investigator# 33418, Minden
  - Site Reference ID/Investigator# 34206, Mittelherwigsdorf
  - Site Reference ID/Investigator# 34219, Moenkeberg
  - Site Reference ID/Investigator# 34216, Mönchengladbach
  - Site Reference ID/Investigator# 53915, Mönchengladbach
  - Site Reference ID/Investigator# 34211, Mönchengladbach
  - Site Reference ID/Investigator# 34214, Mönchengladbach
  - Site Reference ID/Investigator# 53904, Munich
  - Site Reference ID/Investigator# 53956, Munich
  - Site Reference ID/Investigator# 34037, Munich
  - Site Reference ID/Investigator# 53962, Munich
  - Site Reference ID/Investigator# 53912, Munich
  - Site Reference ID/Investigator# 35296, Munich
  - Site Reference ID/Investigator# 53924, Munich
  - Site Reference ID/Investigator# 34041, Munich
  - Site Reference ID/Investigator# 34035, Munich
  - Site Reference ID/Investigator# 34222, Mühlhausen
  - Site Reference ID/Investigator# 34044, Münster
  - Site Reference ID/Investigator# 53970, Münster
  - Site Reference ID/Investigator# 34046, Münster
  - Site Reference ID/Investigator# 34050, Naunhof
  - Site Reference ID/Investigator# 34059, Neubrandenburg
  - Site Reference ID/Investigator# 34062, Neuburg am Inn
  - Site Reference ID/Investigator# 34980, Neunkirchen
  - Site Reference ID/Investigator# 35311, Neuss
  - Site Reference ID/Investigator# 34072, Neustadt
  - Site Reference ID/Investigator# 65630, Neuwied
  - Site Reference ID/Investigator# 82694, Niederbrombach
  - Site Reference ID/Investigator# 34078, Niefern-Öschelbronn
  - Site Reference ID/Investigator# 34081, Nienburg
  - Site Reference ID/Investigator# 34082, Nienburg
  - Site Reference ID/Investigator# 53923, Nuremberg
  - Site Reference ID/Investigator# 34168, Obergünzburg
  - Site Reference ID/Investigator# 34174, Offenburg
  - Site Reference ID/Investigator# 33490, Oldenburg
  - Site Reference ID/Investigator# 53950, Olsberg
  - Site Reference ID/Investigator# 33499, Osnabrück
  - Site Reference ID/Investigator# 54803, Osnabrück
  - Site Reference ID/Investigator# 34715, Ostseebad Damp
  - Site Reference ID/Investigator# 35333, Paderborn
  - Site Reference ID/Investigator# 33503, Papenburg
  - Site Reference ID/Investigator# 33506, Parchim
  - Site Reference ID/Investigator# 33509, Parsberg
  - Site Reference ID/Investigator# 35338, Passau
  - Site Reference ID/Investigator# 33511, Petershagen
  - Site Reference ID/Investigator# 33519, Pinneberg
  - Site Reference ID/Investigator# 33520, Pirna
  - Site Reference ID/Investigator# 33521, Planegg
  - Site Reference ID/Investigator# 33526, Plauen
  - Site Reference ID/Investigator# 33468, Potsdam
  - Site Reference ID/Investigator# 33464, Potsdam
  - Site Reference ID/Investigator# 53940, Pulheim
  - Site Reference ID/Investigator# 33482, Radebeul
  - Site Reference ID/Investigator# 53964, Raststatt
  - Site Reference ID/Investigator# 33485, Ratingen
  - Site Reference ID/Investigator# 35134, Ratingen
  - Site Reference ID/Investigator# 54812, Ratingen
  - Site Reference ID/Investigator# 33888, Regensburg
  - Site Reference ID/Investigator# 33891, Regensburg
  - Site Reference ID/Investigator# 33881, Regensburg
  - Site Reference ID/Investigator# 33884, Regensburg
  - Site Reference ID/Investigator# 53930, Regensburg
  - Site Reference ID/Investigator# 53986, Reichenbach
  - Site Reference ID/Investigator# 53920, Remscheid
  - Site Reference ID/Investigator# 33900, Rendsburg
  - Site Reference ID/Investigator# 33903, Reutlingen
  - Site Reference ID/Investigator# 53982, Rheinfelden
  - Site Reference ID/Investigator# 53908, Rickenbach
  - Site Reference ID/Investigator# 33393, Riesa
  - Site Reference ID/Investigator# 33912, Rinteln
  - Site Reference ID/Investigator# 33921, Rostock
  - Site Reference ID/Investigator# 33929, Rothenburg
  - Site Reference ID/Investigator# 34014, Saarbrücken
  - Site Reference ID/Investigator# 34021, Salzwedel
  - Site Reference ID/Investigator# 53916, Schlangenbad
  - Site Reference ID/Investigator# 34030, Schneeberg
  - Site Reference ID/Investigator# 33550, Schwerin
  - Site Reference ID/Investigator# 35374, Schwerin
  - Site Reference ID/Investigator# 33553, Schwerte
  - Site Reference ID/Investigator# 33557, Seesen
  - Site Reference ID/Investigator# 53944, Siegen
  - Site Reference ID/Investigator# 33565, Sinsheim
  - Site Reference ID/Investigator# 53927, Solingen
  - Site Reference ID/Investigator# 33570, Soltau
  - Site Reference ID/Investigator# 33583, Stadtbergen
  - Site Reference ID/Investigator# 33586, Stadthagen
  - Site Reference ID/Investigator# 53936, Steinhagen
  - Site Reference ID/Investigator# 33602, Stuttgart
  - Site Reference ID/Investigator# 33609, Stuttgart
  - Site Reference ID/Investigator# 33596, Stuttgart
  - Site Reference ID/Investigator# 35387, Suhl
  - Site Reference ID/Investigator# 54808, Tarp
  - Site Reference ID/Investigator# 35433, Thum-Jahnsbach
  - Site Reference ID/Investigator# 53951, Tischenreuth
  - Site Reference ID/Investigator# 33623, Torgelow
  - Site Reference ID/Investigator# 33628, Treuenbrietzen
  - Site Reference ID/Investigator# 53907, Tübingen
  - Site Reference ID/Investigator# 53893, Twistringen
  - Site Reference ID/Investigator# 33635, Ueberlingen-Nussdorf
  - Site Reference ID/Investigator# 53898, Uhlstaedt-Kirchhasel
  - Site Reference ID/Investigator# 33722, Ulm
  - Site Reference ID/Investigator# 65626, Ulm
  - Site Reference ID/Investigator# 33732, Verden an der Aller
  - Site Reference ID/Investigator# 53965, Viersen
  - Site Reference ID/Investigator# 33735, Villingen-Schwenningen
  - Site Reference ID/Investigator# 53914, Vogelsang-Gommern
  - Site Reference ID/Investigator# 53952, Vreden
  - Site Reference ID/Investigator# 54809, Waldbronn
  - Site Reference ID/Investigator# 33740, Waltrop
  - Site Reference ID/Investigator# 34250, Wannsee
  - Site Reference ID/Investigator# 33747, Weener
  - Site Reference ID/Investigator# 53891, Weiden I.d. Oberpfalz
  - Site Reference ID/Investigator# 53921, Weißenfels
  - Site Reference ID/Investigator# 33753, Welzow
  - Site Reference ID/Investigator# 35406, Wiesbaden
  - Site Reference ID/Investigator# 53941, Wiesbaden
  - Site Reference ID/Investigator# 33762, Wiesbaden
  - Site Reference ID/Investigator# 33770, Wilhelmshaven
  - Site Reference ID/Investigator# 53954, Winsen
  - Site Reference ID/Investigator# 53977, Winsen
  - Site Reference ID/Investigator# 33778, Wittlich
  - Site Reference ID/Investigator# 33783, Wolfsburg
  - Site Reference ID/Investigator# 53917, Wuppertal
  - Site Reference ID/Investigator# 35418, Wuppertal
  - Site Reference ID/Investigator# 33716, Würzburg
  - Site Reference ID/Investigator# 33862, Zerbst
  - Site Reference ID/Investigator# 33865, Zeven
  - Site Reference ID/Investigator# 33870, Zwickau
  - Site Reference ID/Investigator# 33878, Zwiesel

REFERENCES:
- [Derived] Behrens F, Koehm M, Schwaneck EC, Schmalzing M, Wittig BM, Gnann H, Greger G, Tony HP, Burkhardt H. Addition or removal of concomitant methotrexate alters adalimumab effectiveness in rheumatoid arthritis but not psoriatic arthritis. Scand J Rheumatol. 2019 Sep;48(5):375-382. doi: 10.1080/03009742.2019.1600717. Epub 2019 Jul 16. PMID 31311386
- [Derived] Scharbatke EC, Behrens F, Schmalzing M, Koehm M, Greger G, Gnann H, Burkhardt H, Tony HP. Association of Improvement in Pain With Therapeutic Response as Determined by Individual Improvement Criteria in Patients With Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2016 Nov;68(11):1607-1615. doi: 10.1002/acr.22884. Epub 2016 Oct 1. PMID 26990995
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rheumatoid Arthritis
Started | 5745
Completed | 1152
Not Completed | 4593
Not completed — Lost to Follow-up | 2363
Not completed — Adverse drug reaction (ADR) | 453
Not completed — Lack of Efficacy | 1193
Not completed — ADR and lack of efficacy | 61
Not completed — Other | 523

BASELINE CHARACTERISTICS:
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 5745
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data available for 5,727 participants
  years | 54.8 (12.8)
Gender [Number; unit: participants] — Gender data missing for 2 participants
  participants
    Female | 4428
    Male | 1315
Region of Enrollment [Number; unit: participants]
  Germany | 5745

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score (DAS) 28
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR), and general health (measured on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10.
  A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: Full analysis set (FAS). Participants with inadequate data or who met other exclusion criteria were not included in the FAS. "n" indicates the number of participants with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
units on a scale
  Month 3 (n=3918) | -1.6 (1.3)
  Month 6 (n=3347) | -1.8 (1.4)
  Month 12 (n=2872) | -2.0 (1.4)
  Month 18 (n=2397) | -2.1 (1.4)
  Month 24 (n=2099) | -2.2 (1.4)
  Month 30 (n=1810) | -2.3 (1.5)
  Month 36 (n=1564) | -2.3 (1.5)
  Month 48 (n=1261) | -2.3 (1.5)
  Month 60 (n=934) | -2.4 (1.5)

2. Primary Outcome: Percentage of Participants in DAS28 Remission
Description: Clinical remission is defined as a DAS28 score of < 2.6. The Disease Activity Score (DAS28) is a validated index of rheumatoid arthritis disease activity calculated from the 28 tender joint count, 28 swollen joint count, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (measured on a visual analog scale [VAS] from 0 to 10 cm). Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
percentage of participants
  Month 3 (n=3918) | 12.8
  Month 6 (n=3347) | 16.9
  Month 12 (n=2872) | 19.4
  Month 18 (n=2397) | 23.0
  Month 24 (n=2099) | 23.3
  Month 30 (n=1810) | 24.3
  Month 36 (n=1564) | 24.0
  Month 48 (n=1261) | 24.7
  Month 60 (n=934) | 25.6

3. Secondary Outcome: Percentage of Participants With a Significant Therapeutic Response
Description: Significant therapeutic response was determined by DAS28 critical difference (Dcrit). A Dcrit response is a statistically determined value that exceeds the threshold of random fluctuation and signifies a positive individual response during treatment. A DAS28-Dcrit individual therapeutic response is defined as a decrease (improvement) in DAS28 from Baseline of ≥ 1.8.
  The Disease Activity Score (DAS28) is a validated index of rheumatoid arthritis disease activity calculated from the 28 tender joint count, 28 swollen joint count, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (measured on a visual analog scale [VAS] from 0 to 10 cm). Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
percentage of participants
  Month 3 (n=3918) | 40.8
  Month 6 (n=3347) | 50.5
  Month 12 (n=2872) | 53.6
  Month 18 (n=2397) | 58.7
  Month 24 (n=2099) | 60.3
  Month 30 (n=1810) | 63.3
  Month 36 (n=1564) | 64.6
  Month 48 (n=1261) | 64.2
  Month 60 (n=934) | 65.5

4. Secondary Outcome: Percentage of Participants With Low, Moderate and High Disease Activity
Description: Low disease activity is defined as a DAS28 score ≤ 3.2; Moderate disease activity as a DAS28 >3.2 to ≤5.1; High disease activity as a DAS28 >5.1.
  The Disease Activity Score (DAS28) is a validated index of rheumatoid arthritis disease activity calculated from the 28 tender joint count, 28 swollen joint count, the erythrocyte sedimentation rate (ESR), and the patient's assessment of global disease activity (measured on a visual analog scale [VAS] from 0 to 10 cm). Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: Full analysis set (FAS) participants with available data at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Month 0: Baseline
- Month 3: 3 months after inclusion
- Month 6: 6 months after inclusion
- Month 12: 12 months after inclusion
- Month 18: 18 months after inclusion
- Month 24: 24 months after inclusion
- Month 30: 30 months after inclusion
- Month 36: 36 months after inclusion
- Month 48: 48 months after inclusion
- Month 60: 60 months after inclusion
Arm/Group | Month 0 | Month 3 | Month 6 | Month 12 | Month 18 | Month 24 | Month 30 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 4400 | 3918 | 3347 | 2872 | 2397 | 2099 | 1810 | 1564 | 1261 | 934
percentage of participants
  Low disease activity | 0.0 | 23.9 | 29.8 | 33.0 | 38.7 | 38.5 | 41.5 | 40.5 | 40.7 | 41.9
  Moderate disease activity | 26.1 | 45.9 | 46.6 | 46.6 | 43.6 | 45.0 | 43.6 | 45.3 | 45.4 | 45.3
  High disease activity | 73.9 | 30.2 | 23.6 | 20.3 | 17.7 | 16.5 | 14.9 | 14.3 | 13.9 | 12.8

5. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Over Time
Description: Erythrocyte sedimentation rate (ESR) indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
mm/hour
  Month 0 (n=4400) | 34.5 (23.1)
  Month 3 (n=4083) | 24.7 (20.4)
  Month 6 (n=3467) | 23.8 (19.9)
  Month 12 (n=2966) | 22.8 (18.9)
  Month 18 (n=2472) | 22.0 (18.4)
  Month 24 (n=2156) | 21.6 (17.7)
  Month 30 (n=1860) | 21.4 (18.1)
  Month 36 (n=1685) | 20.9 (17.5)
  Month 48 (n=1341) | 21.5 (17.8)
  Month 60 (n=998) | 21.2 (17.6)

6. Secondary Outcome: C-Reactive Protein (CRP) Levels Over Time
Description: C-reactive protein (CRP) was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Normal concentration in healthy human serum is usually lower than 10 mg/L, slightly increasing with age.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
mg/L
  Month 0 (n=3852) | 33.7 (63.8)
  Month 3 (n=3209) | 19.8 (56.3)
  Month 6 (n=2671) | 16.1 (29.9)
  Month 12 (n=2192) | 17.0 (89.8)
  Month 18 (n=1770) | 14.9 (68.0)
  Month 24 (n=1573) | 12.3 (27.3)
  Month 30 (n=1355) | 12.0 (26.4)
  Month 36 (n=1211) | 11.0 (22.8)
  Month 48 (n=1000) | 11.6 (27.8)
  Month 60 (n=756) | 9.2 (16.7)

7. Secondary Outcome: Tender Joint Count (TJC) Over Time
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
tender joints
  Month 0 (n=4400) | 12.3 (7.3)
  Month 3 (n=4165) | 6.4 (6.7)
  Month 6 (n=3568) | 5.4 (6.3)
  Month 12 (n=3026) | 4.9 (6.0)
  Month 18 (n=2533) | 4.4 (5.7)
  Month 24 (n=2224) | 4.2 (5.5)
  Month 30 (n=1939) | 4.1 (5.6)
  Month 36 (n=1681) | 4.0 (5.4)
  Month 48 (n=1373) | 3.9 (5.4)
  Month 60 (n=1029) | 3.9 (5.4)

8. Secondary Outcome: Swollen Joint Count (SJC) Over Time
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
swollen joints
  Month 0 (n=4400) | 9.5 (6.3)
  Month 3 (n=4165) | 4.7 (5.3)
  Month 6 (n=3568) | 3.9 (4.9)
  Month 12 (n=3026) | 3.5 (4.5)
  Month 18 (n=2533) | 3.1 (4.3)
  Month 24 (n=2224) | 2.7 (3.9)
  Month 30 (n=1939) | 2.7 (3.9)
  Month 36 (n=1681) | 2.7 (3.8)
  Month 48 (n=1373) | 2.4 (3.8)
  Month 60 (n=1029) | 2.3 (3.6)

9. Secondary Outcome: Hannover Functional Questionnaire (FFbH) Over Time
Description: A self-administered patient questionnaire used to assess patient function based on 18 questions. The numerically coded responses to the questions are added to provide a total patient score. The FFbH was calculated from this patient score by the following formula: FFbH = (patient score x 100) ÷ 2 (number of valid responses). The resulting FFbH score reflects the degree of remaining functional capacity where 0% indicates maximal impairment and 100% indicates maximal functional capacity.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
units on a scale
  Month 0 (n=4360) | 57.7 (23.2)
  Month 3 (n=4075) | 65.1 (23.4)
  Month 6 (n=3498) | 67.1 (23.7)
  Month 12 (n=2978) | 68.3 (23.6)
  Month 18 (n=2493) | 69.4 (23.4)
  Month 24 (n=2194) | 69.9 (23.0)
  Month 30 (n=1908) | 70.1 (23.3)
  Month 36 (n=1715) | 70.4 (23.5)
  Month 48 (n=1394) | 70.0 (23.7)
  Month 60 (n=1048) | 69.9 (24.1)

10. Secondary Outcome: Patients Global Assessment of Disease Activity Over Time
Description: Participants indicated their global assessment of disease activity over the last 7 days on a visual analog scale (VAS) ranging from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
cm
  Month 0 (n=4400) | 6.6 (1.9)
  Month 3 (n=4076) | 4.8 (2.2)
  Month 6 (n=3483) | 4.5 (2.2)
  Month 12 (n=2968) | 4.3 (2.1)
  Month 18 (n=2489) | 4.1 (2.1)
  Month 24 (n=2196) | 4.1 (2.1)
  Month 30 (n=1903) | 4.0 (2.1)
  Month 36 (n=1712) | 3.9 (2.1)
  Month 48 (n=1386) | 3.9 (2.1)
  Month 60 (n=1047) | 3.9 (2.1)

11. Secondary Outcome: Participants Assessment of Pain Over Time
Description: Participants indicated their level of pain over the last 7 days on a visual analog scale (VAS) ranging from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
cm
  Month 0 (n=4388) | 6.8 (2.0)
  Month 3 (n=4079) | 4.7 (2.4)
  Month 6 (n=3484) | 4.3 (2.4)
  Month 12 (n=2966) | 4.1 (2.3)
  Month 18 (n=2491) | 3.9 (2.3)
  Month 24 (n=2190) | 3.9 (2.3)
  Month 30 (n=1904) | 3.8 (2.3)
  Month 36 (n=1712) | 3.7 (2.3)
  Month 48 (n=1383) | 3.8 (2.3)
  Month 60 (n=1048) | 3.7 (2.3)

12. Secondary Outcome: Participants Assessment of Fatigue Over Time
Description: Participants indicated their level of fatigue over the last 7 days on a visual analog scale (VAS) ranging from 0 (best) to 10 (worst) cm; lower scores indicate better patient status.
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
cm
  Month 0 (n=4389) | 6.0 (2.6)
  Month 3 (n=4076) | 4.5 (2.7)
  Month 6 (n=3491) | 4.2 (2.7)
  Month 12 (n=2950) | 4.0 (2.6)
  Month 18 (n=2491) | 3.8 (2.6)
  Month 24 (n=2188) | 3.8 (2.6)
  Month 30 (n=1906) | 3.7 (2.5)
  Month 36 (n=1706) | 3.6 (2.5)
  Month 48 (n=1381) | 3.6 (2.5)
  Month 60 (n=1039) | 3.6 (2.5)

13. Secondary Outcome: Percentage of Participants With Impairment in Daily Activities
Description: Participants were asked to report how many days of impairment in daily activities they had experienced in the last 4 weeks.
Time Frame: Baseline and Months 6, 18, 24, and 30
Population: Full analysis set (FAS) participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Month 0 | Month 6 | Month 18 | Month 24 | Month 30
Number analyzed (Participants) | 4315 | 3428 | 2387 | 2150 | 1860
percentage of participants
  No days of impairment | 17.9 | 38.8 | 45.8 | 44.5 | 45.2
  Less than 7 days of impairment | 28.2 | 34.7 | 33.5 | 35.3 | 36.0
  7 to 14 days of impairment | 28.0 | 16.1 | 13.4 | 13.1 | 12.8
  More than 14 days of impairment | 25.9 | 10.4 | 7.2 | 7.1 | 6.0

14. Secondary Outcome: Number of Days Missed From Work Due to Rheumatoid Arthritis
Description: Participants reported the number of days they had missed from work in the prior 6 months due to rheumatoid arthritis. The Baseline measurement includes data for the prior 12 months.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, 36, 48, and 60
Population: Full analysis set participants who were employed and with available data at each time point (indicated by n)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
days
  Month 0 (n=1503) | 51.0 (78.7)
  Month 6 (n=1173) | 11.6 (35.5)
  Month 12 (n=1016) | 8.6 (30.9)
  Month 18 (n=840) | 6.8 (26.0)
  Month 24 (n=744) | 4.9 (19.8)
  Month 30 (n=637) | 5.2 (19.8)
  Month 36 (n=566) | 5.2 (21.9)
  Month 48 (n=452) | 4.8 (23.6)
  Month 60 (n=339) | 1.8 (9.5)

15. Secondary Outcome: Percentage of Participants With In-patient Hospitalization
Description: The percentage of participants with in-patient hospitalization in the prior 6 months. Baseline data includes in-patient hospitalizations that occurred within the prior 12 months.
Time Frame: Baseline and Months 6, 12, 18, 24, 30, 36, 48, and 60
Population: Full analysis set participants who were employed and with available data at each time point (indicated by n)
Measure: Number; unit: percentage of participants
Arm/Group | Rheumatoid Arthritis
Number analyzed (Participants) | 4400
percentage of participants
  Month 0 (n=4341) | 27.6
  Month 6 (n=3401) | 10.9
  Month 12 (n=2924) | 7.4
  Month 18 (n=2467) | 6.7
  Month 24 (n=2177) | 6.4
  Month 30 (n=1900) | 5.3
  Month 36 (n=1706) | 6.2
  Month 48 (n=1370) | 5.0
  Month 60 (n=1037) | 5.3

16. Secondary Outcome: Percentage of Participants on Concomitant Rheumatoid Arthritis and Pain Relief/Anti-inflammatory Medication
Time Frame: Baseline and Months 3, 6, 12, 18, 24, 30, 36, 48, and 60
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Month 0 | Month 3 | Month 6 | Month 12 | Month 18 | Month 24 | Month 30 | Month 36 | Month 48 | Month 60
Number analyzed (Participants) | 4400 | 4229 | 3611 | 3067 | 2569 | 2250 | 1966 | 1772 | 1435 | 1079
percentage of participants
  Methotrexate | 54.0 | 51.9 | 52.2 | 54.4 | 53.9 | 54.8 | 55.3 | 54.9 | 53.7 | 54.6
  Sulfasalazin | 6.1 | 3.9 | 3.4 | 3.0 | 2.6 | 2.4 | 2.1 | 2.5 | 2.2 | 1.4
  Hydroxychloroquine/Chloroquine | 4.0 | 2.6 | 2.0 | 1.6 | 1.5 | 2.0 | 1.6 | 1.6 | 1.6 | 1.3
  Leflunomide | 20.7 | 15.9 | 13.6 | 13.3 | 12.4 | 11.6 | 11.9 | 10.8 | 9.6 | 8.9
  Other disease-modifying antirheumatic drug | 5.9 | 3.2 | 2.6 | 2.9 | 2.5 | 2.7 | 2.2 | 2.2 | 1.7 | 1.6
  Analgesics | 26.9 | 19.1 | 17.4 | 17.1 | 16.2 | 16.4 | 14.1 | 14.8 | 14.7 | 14.2
  Non-steroidal anti-inflammatory drug | 44.7 | 36.7 | 36.3 | 36.3 | 37.2 | 37.2 | 36.8 | 35.9 | 35.1 | 35.4
  Cyclo-oxygenase 2 (COX-2) Inhibitors | 20.0 | 15.8 | 14.5 | 12.8 | 11.4 | 11.1 | 10.6 | 10.2 | 10.2 | 9.8
  Systemic glucocorticoids | 85.6 | 78.1 | 75.4 | 73.1 | 70.1 | 68.6 | 64.5 | 63.1 | 59.4 | 58.1

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 60-month period.
Arm/Group | Rheumatoid Arthritis
Serious Adverse Events (participants affected / at risk) | 163/5745
Other Adverse Events (participants affected / at risk) | 58/5745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (N=5745)
Pneumonia (Infections and infestations) | 9
Sepsis (Infections and infestations) | 9
Arthritis bacterial (Infections and infestations) | 3
Oral herpes (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Disseminated tuberculosis (Infections and infestations) | 2
Endocarditis (Infections and infestations) | 2
Escherichia sepsis (Infections and infestations) | 2
Fungal infection (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 2
Infection (Infections and infestations) | 2
Papilloma virus infection (Infections and infestations) | 2
Peritoneal tuberculosis (Infections and infestations) | 2
Pneumonia primary atypical (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Abscess limb (Infections and infestations) | 1
Abscess neck (Infections and infestations) | 1
Actinomycosis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Localized infection (Infections and infestations) | 1
Neuroborreliosis (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Pyothorax (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Knee arthroplasty (Surgical and medical procedures) | 7
Surgery (Surgical and medical procedures) | 6
Synovectomy (Surgical and medical procedures) | 4
Foot operation (Surgical and medical procedures) | 3
Arthrodesis (Surgical and medical procedures) | 2
Joint arthroplasty (Surgical and medical procedures) | 2
Skin neoplasm excision (Surgical and medical procedures) | 2
Abscess drainage (Surgical and medical procedures) | 1
Ankle operation (Surgical and medical procedures) | 1
Bone operation (Surgical and medical procedures) | 1
Breast operation (Surgical and medical procedures) | 1
Bursa removal (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Coronary angioplasty (Surgical and medical procedures) | 1
Coronary artery bypass (Surgical and medical procedures) | 1
Hemorrhoid operation (Surgical and medical procedures) | 1
Hip arthroplasty (Surgical and medical procedures) | 1
Hydrocele operation (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Osteosynthesis (Surgical and medical procedures) | 1
Osteotomy (Surgical and medical procedures) | 1
Prostatic operation (Surgical and medical procedures) | 1
Radiotherapy (Surgical and medical procedures) | 1
Renal transplant (Surgical and medical procedures) | 1
Skin graft (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Transurethral incision of prostate (Surgical and medical procedures) | 1
Vertebroplasty (Surgical and medical procedures) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant mesenteric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 5
Impaired healing (General disorders) | 3
Multi-organ failure (General disorders) | 3
Inflammation (General disorders) | 2
Accidental death (General disorders) | 1
Cardiac death (General disorders) | 1
Fat necrosis (General disorders) | 1
Injection site erythema (General disorders) | 1
Injection site swelling (General disorders) | 1
Local swelling (General disorders) | 1
Peripheral edema (General disorders) | 1
Pyrexia (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Coronary artery disease (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 2
Left ventricular failure (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Coronary artery stenosis (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Colitis erosive (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 2
Cerebellar infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Coma (Nervous system disorders) | 1
Hyperkinesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Paresis (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Renal failure acute (Renal and urinary disorders) | 3
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Hepatitis toxic (Hepatobiliary disorders) | 1
Transaminases increased (Investigations) | 2
Catheterization cardiac (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Sleep disorder (Psychiatric disorders) | 2
Decreased activity (Psychiatric disorders) | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Epididymitis (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Dry eye (Eye disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac assistance device user (Social circumstances) | 1
Axillary vein thrombosis (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Subclavian vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rheumatoid Arthritis (N=5745)
Rash (Skin and subcutaneous tissue disorders) | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.